CLINICAL TRIAL: NCT01749709
Title: Effect of Cognitive Stimulation on Recovery After Stroke
Brief Title: Effect of Daily Music Listening on Stroke Recovery
Acronym: MUKU2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Academy of Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 85/180/2011
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Stroke
Keywords: Stroke; Recovery; Music
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Instrumental music listening (Experimental): Daily music listening
  Interventions: Behavioral: Music listening
- Vocal music listening (Experimental): Daily music listening
  Interventions: Behavioral: Music listening
- Audiobook listening (control) (Active Comparator): Daily audiobook listening
  Interventions: Behavioral: Audiobook listening

INTERVENTIONS:
Behavioral: Music listening
  Arms: Instrumental music listening; Vocal music listening
Behavioral: Audiobook listening
  Arms: Audiobook listening (control)

SUMMARY:
Single blind randomized clinical trial including 50 stroke patients to investigate the effect of daily music listening on behavioral, neural and physiological recovery. Patients are randomized (1:1:1) to listen instrumental or vocal music, or audiobooks (recorded book reading) (control). Outcome measures are change in neuropsychological tests, change in self-reported mood, structural and functional magnetic resonance imaging changes and hormonal changes performed at acute, 3-month and 6-month stages.

DETAILED DESCRIPTION:
Please see above

ELIGIBILITY:
Inclusion Criteria:

* Acute Hemispheral stroke

Exclusion Criteria:

* Previous neurological or current psychiatric disease,
* severe aphasia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-12; Primary Completion 2016-04-05 (Actual); Study Completion 2016-04-05 (Actual)

PRIMARY OUTCOMES:
Change in neuropsychological performance (verbal memory) | From acute to 3-month-stage
  Verbal memory summary score (Rivermead Behavioral Memory Test (RBMT) story recall, auditory-verbal learning task)
Change in neuropsychological performance (verbal memory) | From acute to 6-month-stage
  Verbal memory summary score (RBMT story recall, auditory-verbal learning task)

SECONDARY OUTCOMES:
Change in neuropsychological performance (Language skill) | From acute to 3-month-stage
  Verbal fluency task
Change in neuropsychological performance (Language skill) | From acute to 3-month-stage
  Naming test CERAD/Boston Naming Test (BNT)
Change in neuropsychological performance (Language skill) | From acute to 3-month-stage
  Short Token Test
Change in neuropsychological performance (Language skill) | From acute to 6-month-stages
  Verbal fluency task
Change in neuropsychological performance (Language skill) | From acute to 6-month-stages
  Naming test CERAD/BNT
Change in neuropsychological performance (Language skill) | From acute to 6-month-stages
  Short Token Test
Change in mood | From acute to 3-month-stage
  Profile of Mood States
Change in mood | From acute to 6-month-stage
  Profile of Mood States
Change in structural gray matter | From acute to 3-month-stage
  Voxel-based morphometry
Change in structural gray matter changes | From acute to 6-month-stage
  Voxel-based morphometry
Change in structural white matter | From acute to 3-month stage
  Diffusion-weighted imaging
Change in structural white matter | From acute to 6-month stage
  Diffusion-weighted imaging
Change in neuronal function | From acute to 3-month stage
  Resting state/task-based fMRI
Change in neuronal function | From acute to 6-month stage
  Resting state/task-based fMRI
Change in physiological stress level | From acute to 3-month-stage
  Cortisol serum concentration
Change in physiological stress level | From acute to 6-month-stage
  Cortisol serum concentration
Change in physiological stress level | From acute to 3-month-stage
  Beta-endorphin serum concentration
Change in physiological stress level | From acute to 6-month-stage
  Beta-endorphin serum concentration
Change in physiological stress level | From acute to 3-month-stage
  Oxytocin serum concentration
Change in physiological stress level | From acute to 6-month-stage
  Oxytocin serum concentration

CONTACTS AND LOCATIONS:
Overall Officials: Valtteri Kaasinen, MD, Study Chair — Department of Clinical Neurosciences
Locations (1):
- Turku University Hospital, Turku, Finland